CLINICAL TRIAL: NCT00417222
Title: Supplemental Benefit of Angiotensin II Receptor Blocker in Hypertensive Patients With Stable Heart Failure Using Olmesartan (SUPPORT Trial)
Brief Title: Supplemental Benefit of Angiotensin Receptor Blocker in Hypertensive Patients With Stable Heart Failure Using Olmesartan
Acronym: SUPPORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tohoku University (Other)
Responsible Party: Principal Investigator, Hiroaki Shimokawa, MD, PhD, Professor, Tohoku University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-179
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olmesartan medoxomil (Active Comparator): olmesartan medoxomil
  Interventions: Drug: olmesartan medoxomil
- Standard therapy (No Intervention): Standard therapy

INTERVENTIONS:
Drug: olmesartan medoxomil — 5 to 40mg P.O. daily until the end of the study
  Arms: Olmesartan medoxomil

SUMMARY:
The purpose of this study is to investigate whether an angiotensin II receptor blocker (olmesartan), in addition to conventional treatment, will reduce the mortality and morbidity in hypertensive patients with stable chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria.

* Patients with NYHA class II through IV chronic heart failure.
* Patients who have a history of hypertension or those who have antihypertensive medications.
* Patients who are aged 20 years or older and less than 80 years at the entry.
* Stable patients who have angiotensin converting enzyme inhibitor and/or beta-blocker.
* Patients who do not have angiotensin II receptor blocker.

Exclusion Criteria:

* Patients who have renal dysfunction (serum creatinine >=3.0mg/dL) or those who are receiving chronic hemodialysis.
* History of drug hypersensitivity to olmesartan.
* Patients who have severe liver dysfunction.
* History of angioedema.
* History of malignant tumor or life-threatening illness of poor prognosis.
* Pregnant or possibly pregnant patients.
* Cardiovascular surgery within 6months prior to the date of the entry.
* Acute myocardial infarction within 6 months prior to the date of the entry.
* Percutaneous coronary intervention or stent implantation within 6 months prior to the date of the entry.
* Other patients deemed unsuitable as subjects of the study by the treating physician.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2006-11; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
A composite of the following outcomes 1) all-cause death 2) nonfatal acute myocardial infarction 3) nonfatal stroke 4) hospital admission due to congestive heart failure | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.

SECONDARY OUTCOMES:
cardiovascular death | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
death due to heart failure | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
sudden death | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
acute myocardial infarction | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
stroke | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
hospital admission from any cardiovascular reasons | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
fatal arrhythmia or appropriate ICD discharge | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
new-onset diabetes | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
development of renal failure | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
new-onset atrial fibrillation | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
a need to modify treatment procedures for heart failure | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
left ventricular ejection fraction | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.
B-type natriuretic peptide | by the end of the study
  All the patients were enrolled by March, 2010, and were followed-up by the end of March, 2013.

OTHER OUTCOMES:
serum markers for metabolic syndrome | three years
  Blood sampling was performed at the time of and 3 years after randomization. Changes in serum levels of markers for metabolic syndrome (high sensitive C-reactive protein, adiponectin, microRNAs） were examined .

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Shimokawa, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Tohoku University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Tohoku University Graduate School of Medicine, Sendai, Japan

REFERENCES:
- [Derived] Sakata Y, Shiba N, Takahashi J, Miyata S, Nochioka K, Miura M, Takada T, Saga C, Shinozaki T, Sugi M, Nakagawa M, Sekiguchi N, Komaru T, Kato A, Fukuchi M, Nozaki E, Hiramoto T, Inoue K, Goto T, Ohe M, Tamaki K, Ibayashi S, Ishide N, Maruyama Y, Tsuji I, Shimokawa H; SUPPORT Trial Investigators; SUPPORT Trial Investigators. Clinical impacts of additive use of olmesartan in hypertensive patients with chronic heart failure: the supplemental benefit of an angiotensin receptor blocker in hypertensive patients with stable heart failure using olmesartan (SUPPORT) trial. Eur Heart J. 2015 Apr 14;36(15):915-23. doi: 10.1093/eurheartj/ehu504. Epub 2015 Jan 30. PMID 25637937